CLINICAL TRIAL: NCT04064931
Title: Study on Nutritional Deficiencies and Related Factors in Patients With Recurrent Miscarriage
Brief Title: Nutritional Deficiencies About Recurrent Miscarriage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: yuqi2019
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2021-03

CONDITIONS: Abortion, Habitual; Nutritional Status
Keywords: recurrent miscarriage; vitamins
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- recurrent abortion: women of childbearing age who have spontaneous abortion within 20 weeks of pregnancy for 2 or more consecutive times.
  Interventions: Diagnostic Test: Detection of niacin and other vitamins in plasma
- normal pregnancy history: Women of childbearing age who had a normal pregnancy history and are not in pregnancy status now.
  Interventions: Diagnostic Test: Detection of niacin and other vitamins in plasma
- general population: Women of childbearing age in general examination.
  Interventions: Diagnostic Test: Detection of niacin and other vitamins in plasma

INTERVENTIONS:
Diagnostic Test: Detection of niacin and other vitamins in plasma — Detection of niacin and other vitamins in plasma

SUMMARY:
The study plans to recruit patients with recurrent miscarriage and detect their niacin, thiamine, vitamin A, vitamin B6, vitamin B12, vitamin D levels in plasma, evaluating if some lack exists.

DETAILED DESCRIPTION:
Dr. Shi Hongjun from West Lake University has confirmed in a mouse model that a decrease in maternal niacin levels caused by a low niacin diet can lead to stillbirth(HJ Shi, et al. 2017). Due to the lack of a recognized clinical niacin test, it is unclear whether niacin deficiency is associated with abortion. However, some studies have showed: 1. Nearly one-third of pregnant women present low niacin level during the first trimester of pregnancy; 2. Insufficient parent niacin intake is positively correlated with the incidence of congenital heart disease; 3. Vitamin B6 affects niacin metabolism, while maternal B6 deficiency is significantly associated with early abortion. Based on this, the investigators predict that (1) a certain proportion of recurrent abortion women's niacin levels are lower than the normal range of women's normal; (2) supplementation of niacin can reduce the risk of repeated abortion.

There are many methods for detecting niacin, but so far with no reports for large population. Dr. Shi Hongjun from West Lake University used the most sensitive QTRAP 6500+ liquid chromatography tandem mass spectrometer to accurately quantify the concentration of NAD, nicotinamide, niacin and other niacin metabolites in plasma and have optimized the detection process, which would be applicated in this study.

At the same time, studies have shown that pregnant women generally have multiple vitamin deficiency during pregnancy, including plasma thiamine, vitamin A, vitamin B6, vitamin B12 and vitamin D. Therefore, in addition to detecting plasma niacin, this study will also examine the plasma levels of the remaining multivitamins to further explore the impact of nutritional deficiencies on the probability of recurrent miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* Research group 1: Recurrent abortion group: women of childbearing age who have spontaneous abortion within 20 weeks of pregnancy for 2 or more consecutive times.

Control group: 1) Women of childbearing age who had a normal pregnancy history and are not in pregnancy status now. 2) Women of childbearing age in general examination.

Exclusion Criteria:

* patients with confirmed causes unrelated to nutritional deficiencies, including

  1. Both husband and wife have been diagnosed with chromosomal abnormalities or fetal chorionic chromosomal abnormalities;
  2. The patient has been diagnosed with uterine abnormalities;
  3. vaginal bacterial infection or chlamydial infection;
  4. antiphospholipid antibody syndrome;
  5. Other immune system diseases (hypothyroidism, PCOS, hyperprolactinemia);
  6. ovarian function decline (FSH>10mIU/ml);
  7. Cervical insufficiency5.3 Exit criteria:

After being selected, the researcher was withdrawn due to various considerations.

Max Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Recurrent abortion population without confirmed diagnosis of known causes
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Plasma niacin levels in the enrolled population. | 2019-11 to 2020-1

SECONDARY OUTCOMES:
plasma thiamine, vitamin A, vitamin B6, vitamin B12, vitamin D levels of the enrolled population | 2019-11 to 2020-1
full exon sequence of the enrolled population | 2019-11 to 2020-1

CONTACTS AND LOCATIONS:
Overall Officials: Qi Yu, Professor, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Peking Union Medical College and Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The results of outcomes may be presented after the study has been finished.